CLINICAL TRIAL: NCT05436535
Title: Longitudinal Endotyping Of Atopic Dermatitis Through Transcriptomic Skin Analysis (ADRN-12)
Brief Title: Longitudinal Endotyping Of Atopic Dermatitis Through Transcriptomic Skin Analysis
Acronym: LEADS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ADRN-12
Record Dates: First submitted 2022-06-21; First posted 2022-06-29 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab; Triamcinolone Acetonide; Hydrocortisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dupilumab-naïve atopic dermatitis participants (Experimental): On Day 7, dupilumab-naïve AD participants will begin applying topical corticosteroids twice daily to their specified target area, as well as to active lesions on non-target skin.
  Dupilumab-naïve AD participants will return for a Steroid Assessment Visit at Day 35, when response to topical corticosteroids will be evaluated at the target site by TAA and targeted EASI scoring, and overall management of AD body-wide by topical steroid/moisturizer treatment will be evaluated by EASI score.
  Participants who are responsive to topical corticosteroids will continue to use them body-wide through Day 140. Participants who are non-responsive to topical corticosteroids at any time before Day 91 will begin use of dupilumab through their penultimate scheduled visit (Day 140-Day 196) and may continue use of topical corticosteroids outside of their specified target area as needed.
  Interventions: Biological: Dupilumab; Drug: Vanicream- Dupilumab-naïve; Drug: Triamcinolone Acetonide; Drug: Hydrocortisone
- Experienced Dupilumab atopic dermatitis participants (Experimental): AD participants already on dupilumab (for >= 4 months prior to study entry (20 children, 40 adults)) at the start of the study will continue treatment with dupilumab as prescribed by their physician outside of the study. They may also continue treatment with other prescribed topical AD medications outside of the specified target skin area throughout the study; they may continue treatment with other prescribed topical AD medications within the specified target area from Day 7 through Day 140.
  Long-term dupilumab participants will apply Vanicream™ beginning at Day 0 through Day 7. Long-term dupilumab participants will return for assessment visits at Day 63 and 140. At Day 140, participants will resume application of Vanicream™ through the End of Study Assessment (Day 168).
  Interventions: Drug: Vanicream- Experienced Dupilumab
- Non-atopic dermatitis participants (Active Comparator): Approximately 150 will be non-AD controls (including approximately 50 children, 6-17 years of age, and 100 adults, = 18 years of age) Non-AD control participants will apply Vanicream™ beginning at Day 0 through Day 7. Non-AD control participants will return for assessment visits at Day 35, 91, and 140. At Day 140, participants will resume application of Vanicream™ through the End of Study Assessment (Day 168).
  Interventions: Drug: Vanicream- Active

INTERVENTIONS:
Biological: Dupilumab — Adult dupilumab-naïve topical steroid non-responder (EASI >7) participants beginning treatment with dupilumab will initially receive a loading dose of two 300 mg subcutaneous injections. The two injections will be administered at different sites in the abdomen, thighs, or upper arms. Pediatric dupilumab-naïve topical steroid non-responder participants beginning treatment with dupilumab will receive a loading dose, according to their weight. Dupilumab-naïve topical steroid non-responsive participants will continue use of dupilumab on a schedule determined by their age and weight until their penultimate scheduled visit (Day 140-196).
  Other Names: Dupixent
  Arms: Dupilumab-naïve atopic dermatitis participants
Drug: Vanicream- Dupilumab-naïve — Dupilumab-naïve AD participants will apply Vanicream at least twice daily to the specified target skin area over two time periods during the study. First, they will apply starting at Day 0 through Day 7. They will resume application starting at their penultimate visit (Day 140-196) through the End of Study Assessment.
  Arms: Dupilumab-naïve atopic dermatitis participants
Drug: Triamcinolone Acetonide — On Day 7, all dupilumab-naïve AD participants will begin applying triamcinolone 0.1% ointment (provided by the study) twice daily to the specified target area. Additionally, dupilumab-naïve AD participants will apply triamcinolone 0.1% ointment twice daily to active lesions on non-sensitive, non-target skin.
  Between Day 35 and Day 140, dupilumab-naïve AD topical steroid responsive (EASI ≤ 7) participants will apply triamcinolone 0.1% ointment (provided by the study) once or twice daily, per clinician discretion, to the specified target area. Additionally, participants will apply triamcinolone 0.1% ointment once or twice daily, per clinician discretion, to active lesions on non-sensitive skin body wide.
  Between Day 35 and Day 140, dupilumab-naïve topical steroid non-responder (EASI >7) participants may apply triamcinolone 0.1% ointment as needed to active lesions on non-sensitive, non-target skin.
  Arms: Dupilumab-naïve atopic dermatitis participants
Drug: Hydrocortisone — On Day 7, all dupilumab-naïve AD participants will apply hydrocortisone 2.5% ointment twice daily to active lesions on sensitive, non-target skin.
  Between Day 35 and Day 140, dupilumab-naïve AD topical steroid responsive (EASI ≤ 7) participants will apply hydrocortisone 2.5% ointment once or twice daily, per clinician discretion, to active lesions on sensitive skin body wide.
  Between Day 35 and Day 140, dupilumab-naïve topical steroid non-responder (EASI >7) participants may apply hydrocortisone 2.5% ointment as needed to active lesions on sensitive, non-target skin.
  Arms: Dupilumab-naïve atopic dermatitis participants
Drug: Vanicream- Active — Non-AD control participants will apply Vanicream at least twice daily to the specified target skin area over two time periods during the study. First, they will apply starting at Day 0 through Day 7. They will resume application starting at Day 140 through the End of Study Assessment Visit.
  Arms: Non-atopic dermatitis participants
Drug: Vanicream- Experienced Dupilumab — Long-term dupilumab participants will apply Vanicream at least twice daily to the specified target skin area over two time periods during the study. First, they will apply starting at Day 0 through Day 7. They will resume application starting at Day 140 through the End of Study Assessment Visit.
  Arms: Experienced Dupilumab atopic dermatitis participants

SUMMARY:
This is a multi-center, longitudinal study which will characterize the gene expression profiles and transcriptomic endotypes that underlie mild and moderate-severe Atopic dermatitis (AD) and will determine changes in these expression patterns and endotypes in response to standard-of-care treatment. Participants will complete up to ten scheduled study visits with assessment of topical steroid response and dupilumab response (if uncontrolled with topical steroids). Skin samples will be collected at all study visits to determine the gene expression profiles and transcriptomic endotypes that underlie mild vs. moderate-severe AD disease. The investigators will also evaluate the lipidomic, metabolomic, proteomic, and microbiome profiles of AD skin endotypes associated with mild and moderate-severe AD disease. Non-AD participants will serve as a control population.

The primary objective of this study is to determine if the type 2-high non-lesional skin (skin tape) endotype is associated with current mild versus moderate-severe AD disease.

ELIGIBILITY:
Inclusion Criteria:

All Participants:

1. Participant and/or parent guardian must be able to understand and provide informed consent and assent (if applicable)
2. Male or female, 6 years of age or older inclusive at the Screening Visit
3. Participants must agree to apply a stable dose of a study provided topical moisturizer (Vanicream (TM)) at least twice daily between the Baseline Assessment and Day 7 Visits to a specified skin target area
4. Individuals with asthma must adhere to asthma controller medication(s) for the duration of the study
5. Individuals who can become pregnant, as defined in the study manual of procedures, must have a negative pregnancy test at the Baseline Assessment and Day 7 Visits if they do not self-report as pregnant.
6. Individuals who can become pregnant, as defined in the study manual of procedures, must meet either of the following criteria prior to Baseline Assessment:

   1. Willing to remain abstinent from intercourse that may result in pregnancy.
   2. Willing to use Food and Drug Administration (FDA) approved methods of contraception for the duration of the study
7. Participant and/or parent guardian must be able to understand and complete study-related questionnaires.
8. Participants must have adequate sizes of non-lesional skin on extremities or trunk.

   Non-Atopic dermatitis (AD) Participants:
9. No history of AD or food allergy as diagnosed by a physician

   All AD Participants (DNAD and LTD):
10. DNAD and LTD participants must have a history of chronic AD, (according to the Atopic Dermatitis Research Network [ADRN] Standard Diagnostic Criteria [Appendix B]), that has been present for at least 1 year before the Screening Visit.
11. Must agree to refrain from applying topical steroid to a specified target area between the Baseline Assessment and Day 7 Visit

    DNAD Participants:
12. DNAD participants must have active lesions on the upper or lower extremities or trunk of sufficient size and in the required locations, as specified in the study manual of procedures (MOP), for specimen collection at the Baseline Assessment and Steroid Initiation (Day 7) Visits.

    LTD Participants:
13. Long-term dupilumab participants must be currently receiving dupilumab and must have started dupilumab treatment >= 4 months prior to the Screening Visit

Exclusion Criteria:

1. Inability or unwillingness of a participant or parent guardian to comply with study protocol
2. Have a genetic relative (e.g., parent, sibling, grandchild, half-sibling) or household member (e.g., spouse) already enrolled in the study
3. Weight less than 15 kg
4. Known systemic hypersensitivity to any of the excipients of the study treatments (Vanicream (TM), hydrocortisone, triamcinolone, or dupilumab)
5. Have any skin disease other than Atopic dermatitis (AD) that might compromise the stratum corneum barrier (e.g., bullous diseases, psoriasis, cutaneous T cell lymphoma [also called Mycosis Fungoides or Sezary syndrome], dermatitis herpetiformis, Hailey-Hailey, or Darier's disease)
6. Known or suspected immunosuppression, including history of invasive opportunistic infections (e.g. tuberculosis, histoplasmosis, listeriosis, coccidioidomycosis, pneumocystis, aspergillosis) despite infection resolution, or otherwise recurrent immune-compromised status, as judged by investigator
7. Known history of human immunodeficiency virus (HIV) infection
8. Ocular disorder that in the opinion of the investigator could adversely affect the individual's risk for study participation. Examples include, but are not limited to, individuals with a history of or active case of herpes keratitis; Sjogren's Syndrome, Keratoconjunctivitis Sicca, or Dry Eye Syndrome that require daily use of supplemental lubrication; or individuals with ocular conditions that require the regular use of ocular corticosteroids or cyclosporine
9. Parasitic infection, except for vaginal trichomoniasis, within 12 months of the Screening Visit, or high risk for contracting parasitic infections (e.g. living in or traveling to endemic areas)
10. History of malignancy within 5 years before the Screening Visit (completely treated in situ carcinoma of the cervix, and completely treated and resolved non-metastatic squamous or basal cell carcinoma of the skin or melanoma in situ are not exclusionary)
11. History of non-malignant lymphoproliferative disorders
12. History of alcohol or drug abuse within 2 years before the Screening Visit
13. History of keloid formation (exclusionary for adult participants only)
14. History of hypersensitivity to local anesthetics (e.g., lidocaine or Novocain), bleeding disorders, or treatment with anticoagulants or other conditions in adult participants that would make the biopsy procedure inadvisable
15. History of serious life-threatening reaction to tape or adhesives
16. Individuals with asthma who have required use of a systemic corticosteroid within 3 months prior to the Baseline Assessment Visit or who require a dose greater than 880 mcg/day of fluticasone propionate or equivalent inhaled corticosteroid to maintain asthma control.
17. Planned major surgical procedure during study participation that could affect study participation or outcome assessment, per PI discretion
18. Chronic or acute infection requiring treatment with systemic antibiotics, antivirals, antiparasitics, antiprotozoals, or antifungals within 4 weeks before the Baseline Assessment Visit, or superficial skin infection within 1 week before the Baseline Assessment Visit
19. Pregnant or breast-feeding women, or women planning to become pregnant or breastfeed during the study
20. Use of any systemic (oral, intravenous (IV), intramuscular (IM)) immunosuppressive/immunomodulating therapies (e.g. steroids, cyclosporine, Janus kinase inhibitors, mycophenolate, azathioprine, or methotrexate) within 4 Weeks of the Baseline Assessment Visit, or any condition that, in the opinion of the investigator, will likely require such treatment(s) during study participation
21. Treatment with biologics (other than dupilumab) as follows:

    1. Any cell-depleting agents, including but not limited to rituximab, within 6 months before the Baseline Assessment Visit, or until lymphocyte and CD 19+ lymphocyte count returns to normal, whichever is longer
    2. Omalizumab, Infliximab, adalimumab, golimumab, certolizumab pegol, abatacept, etanercept, anakinra within 16 weeks before the Baseline Assessment Visit for any indication
    3. Other biologics within 5 half-lives (if known) or 16 weeks before the Baseline Assessment Visit, whichever is longer
22. Treatment with a live (attenuated) vaccine within 7 weeks before the Baseline Assessment Visit or planning to receive a live vaccine during the study
23. Ongoing participation in another research study involving any of the following:

    1. Current or planned use of an investigational drug or device.
    2. Current or planned use of prohibited medications or procedures
    3. Substantial time commitment and/or study requirements that may interfere with the participant's ability to comply with LEADS study requirements
24. Use of investigational drug within 8 weeks or within 5 half-lives (if known), whichever is longer, before the Baseline Assessment Visit
25. Use of topical calcineurin inhibitors (tacrolimus or pimecrolimus), topical phosphodiesterase inhibitors (crisaborale), or topical JAK inhibitors (ruxolitinib) within 1 week before the Baseline Assessment Visit
26. Use of phototherapy (such as narrowband ultraviolet B [NBUVB], ultraviolet B [UVB], ultraviolet A1 [UVA1], psoralen + UVA [PUVA]) or a tanning booth/parlor within 4 weeks of the Baseline Assessment Visit.
27. Treatment with bleach bath within 1 week before the Baseline Assessment Visit
28. Use of a chlorinated hot tub within 1 week before the Baseline Assessment Visit
29. Initiation of treatment with prescription moisturizers or moisturizers containing ceramide, hyaluronic acid, urea, or filaggrin (FLG) during the study period (participants may continue using stable doses of such moisturizers on body areas other than the target area if initiated before the Baseline Assessment Visit)

    1. Participants may continue using stable doses of such moisturizers on body areas other than the target area if initiated before the Baseline Assessment.
    2. Initiation of prescription moisturizer is not exclusionary when only applied to the face, neck, palms, or soles.
30. Planned or anticipated use of any prohibited medications or procedures during study participation.
31. Past or current medical problems or findings from physical examination that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2025-04-07 (Actual); Study Completion 2025-10-24 (Actual)

PRIMARY OUTCOMES:
Mild (EASI ≤ 7) vs. moderate-to-severe (EASI > 7) AD severity between type 2-high vs. type 2-low endotype from non-lesional skin transcriptome in the dupilumab-naïve AD adults and children. | At Day 7
  Eczema Area and Severity Index (EASI) is a composite score (range: 0-72) measuring physical signs of atopic dermatitis (AD), including area of involvement and severity. Severity components include erythema, papulation, excoriation and lichenification [0=absent, 1=mild, 2=moderate, 3=severe] for each body region (head/neck, trunk, arms, legs). Area of involvement (%) is assessed for each body region. Area and severity of each body region is weighted based on size of region, and region scores are added for the total score. Scores ≤7 are considered mild AD severity, >7 are considered moderate-to-severe.

SECONDARY OUTCOMES:
Normalized gene counts expressed in non-lesional skin transcriptome between non-AD vs. mild dupilumab-naïve AD adults and children. | At Day 7 and Days 168-224 (End of Study)
  Gene counts are produced by whole transcriptome sequencing (WTS) on the non-lesional skin tape strips collected at Day 7 and Day 168-224 (End of Study). These counts are then normalized by variance stabilizing transformation (VST).
Normalized gene counts expressed in non-lesional skin transcriptome between non-AD vs. moderate-to-severe dupilumab-naïve AD adults and children. | At Day 7 and Days 168-224 (End of Study)
  Gene counts are produced by whole transcriptome sequencing (WTS) on the non-lesional skin tape strips collected at Day 7 and Day 168-224 (End of Study). These counts are then normalized by variance stabilizing transformation (VST).
Change in normalized gene counts expressed in non-lesional skin transcriptome from Day 7 to Day 168-224 among Non-AD, Topical Steroid Responders, Dupilumab Responders, Dupilumab Non-Responders, and Long-term Dupilumab AD adults and children. | At Day 7 and Days 168-224 (End of Study)
  Gene counts are produced by whole transcriptome sequencing (WTS) on the non-lesional skin tape strips collected at Day 7 and Day 168-224 (End of Study). These counts are then normalized by variance stabilizing transformation (VST). The change in normalized gene counts is calculated from Day 7 to Day 168-224 (End of Study) within each group.

CONTACTS AND LOCATIONS:
Overall Officials: Donald Leung, M.D., Ph.D., Study Chair — National Jewish Health: Division of Pediatric Allergy and Clinical Immunology; Max A. Seibold, Ph.D., Study Chair — National Jewish Health: Division of Pediatric Allergy and Clinical Immunology
Locations (10):
- United States (10):
  - University of California, San Diego: Dermatology Clinical Trials Unit, La Jolla, California
  - Children's Hospital Los Angeles: Division of Clinical Immunology & Allergy, Los Angeles, California
  - National Jewish Health: Division of Pediatric Allergy and Clinical Immunology, Denver, Colorado
  - Boston Children's Hospital: Department of Immunology, Boston, Massachusetts
  - Icahn School of Medicine at Mount Sinai: Department of Pediatrics Allergy & Immunology, New York, New York
  - University of Rochester Medical Center: Department of Dermatology, Rochester, New York
  - North Carolina Children's Hospital: Department of Pediatrics, Division of Allergy, Immunology and Rheumatology, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital Medical Center: Asthma Center, Cincinnati, Ohio
  - Oregon Health & Science University: Department of Dermatology, Portland, Oregon
  - University of Pennsylvania, Perelman Center for Advanced Medicine: Department of Dermatology, Philadelphia, Pennsylvania

REFERENCES:
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — http://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — http://www.niaid.nih.gov/